CLINICAL TRIAL: NCT05871762
Title: Choice of the Optimal Treatment Strategies for Mid-low REctal Cancer-a National Multi-center, Prospective, Real World Study
Brief Title: Choice of the Optimal Treatment Strategies for Mid-low REctal Cancer
Acronym: COMREC
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-PUMCH-C-027
Record Dates: First submitted 2023-05-10; First posted 2023-05-23 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Registry study, no specific intervention — Registry study, no specific intervention

SUMMARY:
The purpose of this study is to compare the efficacy, prognosis, health economics of different treatment modalities of mid-low rectal cancer in different centers in China, and to conduct cost utility analysis (CUA) on the treatment process of rectal cancer to explore the best treatment modality that meets the actual need of medical units in each region and at each level. The investigators hope to provide evidence-based medical suggestions for medical quality control of rectal cancer and revision of clinical guidelines, and provides a source of decision making for medical management and medical insurance.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed rectal adenocarcinoma
* located within 12cm below the anal verge

Exclusion Criteria:

* diagnosed with distant metastasis
* multiple primary colorectal cancers
* history of previous malignant tumors
* Pregnant or lactating women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: mid-low rectal cancer patients
Sampling Method: Probability Sample
Enrollment: 3705 (Estimated)
Dates: Start 2023-06-04 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
3-year OS | 3 years
  3-year overall survival

SECONDARY OUTCOMES:
3-year DFS | 3 years
  3-year disease-free survival
3-year LR | 3 years
  3-year local recurrence rate
3-year distant metastasis rate | 3 years
  3-year distant metastasis rate
neoadjuvant therapy rate | at the time point of surgery of the primary lesion
  the percentage of patients who underwent standard neoadjuvant therapy
adjuvant therapy rate | at the time point of 3-year follow up
  the percentage of patients who underwent standard adjuvant therapy
EUS/MRI assessment rate | at the time point of surgery of the primary lesion
  the percentage of patients who underwent standard rectal EUS/MRI assessment
R0 resection rate | at the time point of surgery of the primary lesion
  the percentage of patients who underwent R0 resection
CCR | immediately after the completion of neoadjuvant therapy assessment
  Clinical Complete Response
pCR | immediately after the completion of surgery
  Pathologic Complete Response
30-day mortality | 30 days after the surgery
  death occurring within 30 days of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China